CLINICAL TRIAL: NCT06875869
Title: Comparative Effects of Jones and Ischemic Compression Technique on Pain, Range of Motion and Disability in Patients With Cervicogenic Headache
Brief Title: Ischemic Compression Technique Versus Jones Technique in Cervicogenic Headache Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0152
Record Dates: First submitted 2025-03-10; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Cervicogenic Headache
Keywords: Cervicogenic headache; Disability evaluation; Ischemic compression therapy; Pain assessment; Range of motion; Trigger point
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-A (Jones technique) (Experimental): Patients will receive Jones technique for the Sternocleidomastoid and upper fibers of Trapezius.
  Interventions: Other: Jones technique
- Group-B (Ischemic compression therapy) (Active Comparator): Patients will receive Ischemic compression for the Sternocleidomastoid and upper fibers of Trapezius
  Interventions: Other: Ischemic compression therapy

INTERVENTIONS:
Other: Jones technique — In the Jones technique, pressure will be applied on the tender point and the patient's head will be flexed laterally to the side of the tender point, followed by a shoulder abduction of approximately 90 degrees. This position will be held for 90 s and then patient position will be passively returned to the initial position. This will be repeated three times in each session. Patients will receive two treatment sessions per week for 6 weeks
  Arms: Group-A (Jones technique)
Other: Ischemic compression therapy — Patients will receive ischemic compression of the trigger points of the upper trapezius and sternocleidomastoid muscle with hold time varying between 30 seconds to 1 minute repeated 3 to 5 times in each session. Patients will receive two treatment sessions per week for 6 weeks
  Arms: Group-B (Ischemic compression therapy)

SUMMARY:
The primary objective of the study is to determine the effects of Jones and Ischemic compression technique on pain, range of motion and disability in patients with cervicogenic headache. Cervicogenic headache is a distinctive type of secondary headache where the pain originates from structures in the neck or cervical spine and radiates to the head. Trigger point release has been associated with decrease in symptoms of patients with cervicogenic headache. This study will be a randomized clinical trial with the sample size of 32 patients. Participants will be randomly allocated into two groups: Group A and Group B. The setting of the study will be Bahawal Victoria Hospital, Bahawalpur. Group A will receive Jones technique of trigger points of the upper trapezius and sternocleidomastoid muscle while Group B will receive ischemic compression of the trigger points of the upper trapezius and sternocleidomastoid muscle. Patients of both groups will receive two treatment sessions per week for 6 weeks. Both groups will receive hot pack for 10 minutes, TENS for 15 minutes and strengthening exercises for deep neck flexors (chin tuck and head raise with ten repetitions of 10-second duration, with a 10-second rest interval between each contraction) as baseline treatment protocol. NPRS, HDI and FRT will be used as outcome measure tools. Data will be analyzed using SPSS version 25.0 with the p-value of <0.05 taken as significant difference.

DETAILED DESCRIPTION:
Cervicogenic headache (CGH) is a secondary headache caused by a disorder of the cervical spine and its disc or bony and/or periarticular components and is often accompanied by neck pain The prevalence cervicogenic headache of in the general population has been reported to be 2.2%-4.1% and appears to predominate in women four times more than in men. Noninvasive treatment techniques consist mainly of electrotherapy, manual therapy (MT), and exercise prescription. Myofascial Trigger Point (MTrP) activity is one of the leading causes of CGH. Jones technique and Ischemic compression ( IC) are two treatment options for trigger points. Cervicogenic headaches are a growing problem impacting daily life, research on cervicogenic headaches is crucial to understand the link between neck issues and headaches, and develop more effective long-term treatment options. In view of the above, the current study aims to evaluate the effectiveness of Physiotherapy interventions i.e. Jones and Ischemic compression technique for Myofascial Trigger Points (MTrPs) of Sternocleidomastoid and upper Trapezius in treating cervicogenic headache.

The current study will help us in determining whether use of these techniques has any significant advantage over conventional treatment for pan and disability in CGH patients. Understanding the most effective therapeutic approach can guide practitioners in selecting evidence-based interventions, ultimately improving the overall well-being of patients suffering from cervicogenic headache.

ELIGIBILITY:
Inclusion Criteria:

* Both males and females
* 25-35 years of age
* Individuals satisfying the Cervicogenic Headache criteria
* Positive Simon's criteria for trigger points

Exclusion Criteria:

* primary headaches (i.e., migraine, tension type headache)
* bilateral headache
* Presence of any red flags
* cervical spinal stenosis
* evidence of central nervous system involvement
* prior surgery to the head or neck

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2025-09-02 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 6 weeks
  It is a standardized self-reporting scale consisting of a horizontal line used to estimate the subjective level of pain intensity. It is a 11 point numerical scale, corresponding to the degree of pain. 0= no pain, 1-2-3 = mild pain, 4-5-6 = moderate pain, 7-8-9-10 = severe pain. The patients will be asked to select from that 11 points numerical continuum the number that corresponds to their perceived pain intensity
Headache Disability index (HDI) | 6 weeks
  This scale is intended to help discover impact of headache. It contains 27 questions in total. First two questions are about frequency of headache and remaining 25 regarding impact of headache on daily life of the person. Each question has three possible answers. "yes " will score 4 points, " sometimes" will score 2 and "no" will give 0 score. A total score of 10 - 28 is regarded as an indicator of light disability, the score of 30-48 represents moderate disability, 50-68 expresses severe disability, and 72 or above marks complete disability
Flexion Rotation test (FRT) | 6 weeks
  Flexion rotation test is used to measure cervical range of motion employing a goniometer. Impairment in upper cervical spine mobility is associated with cervicogenic headache severity and disability. Measures of such mobility include the flexion-rotation test (FRT), which requires full cervical flexion and may be influenced by lower cervical spine dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Ghulam Fatima, PHD*, Principal Investigator — Riphah International University
Locations (1):
- Bahaval Victoria Hospital, Bahawalpur, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Page P. Cervicogenic headaches: an evidence-led approach to clinical management. Int J Sports Phys Ther. 2011 Sep;6(3):254-66. PMID 22034615
- [Background] Knackstedt H, Bansevicius D, Aaseth K, Grande RB, Lundqvist C, Russell MB. Cervicogenic headache in the general population: the Akershus study of chronic headache. Cephalalgia. 2010 Dec;30(12):1468-76. doi: 10.1177/0333102410368442. Epub 2010 May 19. PMID 20974607
- [Background] Bogduk N, Govind J. Cervicogenic headache: an assessment of the evidence on clinical diagnosis, invasive tests, and treatment. Lancet Neurol. 2009 Oct;8(10):959-68. doi: 10.1016/S1474-4422(09)70209-1. PMID 19747657
- [Background] Garcia JD, Arnold S, Tetley K, Voight K, Frank RA. Mobilization and Manipulation of the Cervical Spine in Patients with Cervicogenic Headache: Any Scientific Evidence? Front Neurol. 2016 Mar 21;7:40. doi: 10.3389/fneur.2016.00040. eCollection 2016. PMID 27047446
- [Background] Olesen J. International Classification of Headache Disorders. Lancet Neurol. 2018 May;17(5):396-397. doi: 10.1016/S1474-4422(18)30085-1. Epub 2018 Mar 14. No abstract available. PMID 29550365